**PRINCIPAL INVESTIGATOR:** Fatima Karzai, M.D.

STUDY TITLE: Neoadjuvant Androgen Deprivation and Enzalutamide:

Using Multiparametric MRI to Evaluate Intraprostatic Tumor Responses and Androgen Resistance Patterns in Newly

Diagnosed Prostate Cancer

STUDY SITE: NIH Clinical Center

Cohort: Standard

Consent Version: *05/16/2022* 

#### WHO DO YOU CONTACT ABOUT THIS STUDY?

**Principal Investigator:** Fatima Karzai, M.D.

Phone: 301-480-7174

Email: fatima.karzai@nih.gov

This consent form describes a research study and is designed to help you decide if you would like to be a part of the research study.

The remaining document will now describe the research study in more detail. This information should be considered before you make your choice. Members of the study team will talk with you about the information in this document. Some people have personal, religious, or ethical beliefs that may limit the kinds of medical or research interventions in which they would want to participate. Take the time you need to ask any questions and discuss this study with NIH staff, and with your family, friends, and personal health care providers.

If the individual being asked to participate in this research study is not able to give consent for themselves, you, as the Legally Authorized Representative, will be their decision-maker and you are being asked to give permission for this person to be in this study. For the remainder of this document, the term "you" refers to you as the decision-maker and/or the individual being asked to participate in this research.

#### IT IS YOUR CHOICE TO TAKE PART IN THE STUDY

You may choose not to take part in this study for any reason. If you join this study, you may change your mind and stop participating in the study at any time and for any reason. In either case, you will not lose any benefits to which you are otherwise entitled. However, to be seen at the NIH, you must be taking part in a study or are being considered for a study. If you do choose to leave the study, please inform your study team to ensure a safe withdrawal from the research.

#### WHY IS THIS STUDY BEING DONE?

This study is being done to develop improved techniques for the detection of prostate cancer both before and after pre-operative treatment. In this study we will be testing whether we can use a

### PATIENT IDENTIFICATION

**Consent to Participate in a Clinical Research Study** 

NIH-2977 (4-17)

File in Section 4: Protocol Consent (1)

Version Date: 05/16/2022


technique called multi parametric magnetic resonance imaging (mpMRI) for localizing and detecting prostate cancer. We also want to determine if two drugs used in combination prior to surgery will provide any benefit to people who have non-metastatic prostate cancer (cancer that has not spread to other parts of the body). There are several therapies available to treat prostate cancer. This study will utilize a combination of androgen deprivation therapy (example goserelin or leuprolide) and enzalutamide followed by surgery. Goserelin and enzalutamide are both approved by the Food and Drug Administration (FDA) to treat prostate cancer. However, less is known about the effect of using these drugs in combination before surgery.

## Why are you being asked to take part in this study?

You are being asked to take part in this study because you have been recently diagnosed with prostate cancer that is non-metastatic and you are a candidate for a radical prostatectomy following treatment. After considering all treatment options discussed with you, including possible radiation therapy options, you have decided to undergo a radical prostatectomy as part of the standard care for your cancer.

## How many people will take part in this study?

About 55 people at NIH will take part in this study.

## **Description of Research Study**

### What will happen if you take part in this research study?

### Before you begin the study

Certain standards (criteria) have been established to ensure that you are a medically appropriate candidate for this trial. These criteria also make sure that the results of this study can be used to help make decisions about treating other patients. We will record your medical history and give you a physical examination. You will undergo standard blood tests including a complete blood count, chemistry panel, and prostate-specific antigen (PSA) levels, and scans and x-rays as part of the NCI Screening Protocol.

#### **During the study**

If you are found to be eligible for this trial, you will be asked to complete the following tests and procedures:

- Physical Exam and vital signs monthly
- Provide samples of blood and urine for standard and research testing. The total amount of blood we will draw for research in this study is about 75ml (5 tablespoons).
- ECG before treatment and surgery
- 3T mpMRI after 6 months of treatment

You will be offered the opportunity to fill in your wishes for research and care, and assign a substitute decision maker on the "NIH Advance Directive for Health Care and Medical Research Participation" form so that another person can make decisions about your medical care in the event that you lose the ability to provide on-going consent during the course of the study.

3T mpMRI

#### PATIENT IDENTIFICATION

### **Consent to Participate in a Clinical Research Study**

NIH-2977 (4-17)

File in Section 4: Protocol Consent (1)


During the procedure, you will be asked to lie down on the MRI platform and turn on your side with your back to the nurse or technician. A brief digital exam will be performed to assess the anus for safe probe insertion and then an endorectal probe will be inserted. Then, you will need to turn on your back so that you can be positioned within the bore of the scanner. You will also be given earphones or earplugs to help block out noise from the MRI scanner.

While inside the MRI bore and during the course of the scan, you, doctors, and technologists may communicate via a microphone and room loudspeaker system. In order for us to obtain the best images and data, you will need to remain motionless and relaxed during the entire exam, which lasts about 60 minutes.

Upon completion of the exam, you will be moved outside of the MRI bore and the endorectal probe will be removed.

Following these tests and procedures you will take the two study medications for 6 months. Enzalutamide is given by mouth. You will take 4 pills one time per day. Goserelin is given by injection once every 3 months for 6 months (2 doses in 6 months). If Goserelin is not available another form of androgen deprivation therapy may be prescribed. The doses and how you take these alternate medications may be different. If an alternate medication is prescribed, the study staff will let you know how much medication and how often you will need to take it.

You will be asked to return to the clinic once each month for safety tests which will include a physical exam, having your vital signs taken and standard blood tests.

If your PSA rises during the study, other treatment options may be available to you including new imaging studies, re-biopsy and possibly earlier surgery. The study doctor will discuss all these options with you and you will have the opportunity to decide which is best for your care.

### Research Studies

Tumor samples that have been collected during surgery will be analyzed by the pathologist and the results will be discussed with you.

All of your samples collected for research purposes on this study (such as your tumor, urine and blood) may be used to look for specific changes in the DNA of genes that may cause prostate cancer or other types of cancer. DNA (also called deoxyribonucleic acid) in the cells carries genetic information and passes it from one generation of cells to the next – like an instruction manual. Normal tissue contains the DNA (instructions) that you were born with, DNA in tumor cells has changed – or mutated – and we think that change in the DNA is what causes tumors to form and to grow.

To look at your DNA, we may use do what is called "whole genome sequencing." This is where we will do special tests in the lab to look at the entire sequence, or order, of how your DNA is put together. This is what makes you unique.

To determine which parts of the DNA have mutated, we will compare the DNA in your tumor cells to DNA from your normal cells. We will then analyze the results from similar tumors to see if there are any changes in the DNA that are common to a particular type of tumor. To examine your tissue we may use several different techniques depending on the type of tissue we collect. These could include growing cell lines (cells which keep dividing and growing in the laboratory, sometimes for years allowing us to continually study those cells), xenograft studies (placing or

### PATIENT IDENTIFICATION

Consent to Participate in a Clinical Research Study

NIH-2977 (4-17)

File in Section 4: Protocol Consent (1)


Page **3** of **14** 

growing cells in another animal, such as mice), and looking in detail at the parts of the genes that produce specific proteins.

However, you should know that the analyses that we perform in our laboratory are for research purposes only; they are not nearly as sensitive as the tests that are performed in a laboratory that is certified to perform genetic testing or testing for routine clinical care. For these reasons, we will not give you the results of the research tests done on your research samples in most cases. There may be exceptions to what we share with you and this is described in the next section, "Return of research results."

#### Return of research results

When we are examining your DNA, it is possible that we could identify possible changes in other parts of your DNA that are not related to this research. These are known as "incidental medical findings".

#### These include:

- Changes in genes that are related to diseases other than cancer
- Changes in genes that are not known to cause any disease. These are known as normal variations.
- Changes in genes that are new and of uncertain clinical importance. This means that we do not know if they could cause or contribute to a disease or if they are normal variations.

Since the analyses that we perform in our laboratory are not nearly as sensitive as the tests that are performed in a laboratory that is certified to perform genetic testing, the genetic changes that we find may or may not be valid. Therefore, we do not plan to inform you of all of the genetic results of testing on your tissue and blood that is performed in our research lab. However, in the unlikely event that we discover a finding believed to be clinically important based on medical standards at the time we first analyze your results, we will contact you. This could be many years in the future. We will ask you to have an additional tube of blood drawn to verify the findings we have seen in our lab. If the results are verified, you will be re-contacted and offered a referral to a genetic healthcare provider to discuss the results.

Note: In order for us to contact you about genetic variants as described above, we must maintain your up to date contact information. This will allow us to contact you at the time findings are discovered.

### When you are finished taking the drugs

After you have completed the study medications, you will be asked to undergo another 3T mpMRI, blood tests and then you will have surgery to remove your prostate. This surgery may be performed at either the Clinical Center or Walter Reed Bethesda. After the surgery you will return for a follow up visit about 6-10 weeks after your prostate is removed and then we will call you yearly for the next five years to check your PSA level. PSA levels may be obtained at NIH or through a local provider.

PATIENT IDENTIFICATION

Consent to Participate in a Clinical Research Study

NIH-2977 (4-17)

File in Section 4: Protocol Consent (1)


#### **Standard of Care Treatment**

Treatments covered under this study include a combination of medications and surgery to treat your cancer. These treatments will not be experimental. Your doctors will describe your treatment plan to you in detail before asking you to sign this consent form. You may be asked to sign a separate consent form for any treatment procedures not outlined in this consent.

#### **Birth Control**

If you are the partner of a woman who can become pregnant, you and your partner will need to practice an effective form of birth control before starting study treatment, during study treatment, and for 3 months after you finish study treatment. If you think that your partner is pregnant, you should tell your study doctor or nurse at once.

Effective forms of birth control include:

- abstinence
- intrauterine device (IUD)
- hormonal [birth control pills, injections, or implants]
- tubal ligation
- vasectomy

### **Risks or Discomforts of Participation**

## What side effects or risks can I expect from being in this study?

As with all treatments, there are several side effects or risks from the treatments provided in this study. However, doctors don't know all the side effects that may happen with this combination of drugs, so it is important to report any changes that you notice, even if your study team does not ask specifically about them. Side effects may be mild or severe. Your study team will give you medicines to help lessen side effects. Many side effects go away with those medicines and others may go away soon after you stop treatment. In some cases, side effects can be serious, long-lasting, or may never go away. In very rare instances, they could cause death.

#### Possible side effects of enzalutamide:

| Likely | Less Likely | Rare but Serious |
|---|---|---|
| <ul> <li>Ankle swelling</li> <li>Fatigue</li> <li>Headache</li> <li>Hot flashes</li> <li>Diarrhea</li> <li>Low blood counts</li> <li>Back pain</li> <li>Upper respiratory tract infection</li> <li>Nipple tenderness</li> </ul> | <ul> <li>High blood pressure</li> <li>Dizziness, anxiety</li> <li>Dry skin</li> <li>Blood in urine</li> <li>Jaundice</li> <li>Weakness of muscles</li> </ul> | • Seizures |

#### PATIENT IDENTIFICATION

Consent to Participate in a Clinical Research Study

NIH-2977 (4-17)

File in Section 4: Protocol Consent (1)


## Possible Side effects of goserelin:

| Likely (greater than 5%) | Less Likely (1%–5%) | Rare but Serious |
|---|---|---|
| <ul> <li>Hot flashes</li> <li>Generalized pain or pain in the pelvis or bone</li> <li>Enlarged breasts</li> <li>Weakness</li> </ul> | <ul> <li>Pain in abdomen and/or back</li> <li>Flu-like symptoms</li> <li>Headache</li> <li>Cardiac problems (chest pain, clots, varicose veins)</li> <li>Diarrhea</li> <li>Vomiting blood</li> <li>Sugar in blood</li> <li>Low red cells (anemia)</li> <li>Swelling in hands or feet</li> <li>Dizziness</li> <li>Numbness or tingling</li> <li>Frequent urination, unable to void, unable to hold urine, urinary infection, blood in urine</li> <li>Impotence</li> <li>Itchy skin</li> <li>Herpesvirus of the skin</li> </ul> | <ul> <li>Infection in blood</li> <li>Heart failure</li> <li>Stroke</li> <li>Clot that may travel to lungs or brain</li> </ul> |

#### Other Risks

### **ECG**

There are no significant risks or discomforts associated with an ECG. Some patches will be adhered to your skin that may cause some reddening or slight itching.

#### Blood draws

There may be some side effects associated with the procedures for drawing blood in this study, but the person drawing your blood will attempt to minimize this discomfort. Side effects include pain and bruising in the area where the needle is inserted, lightheadedness, and rarely, fainting. When large amounts of blood are collected, low red blood cell count (anemia) is a risk.

#### Urine collection

There are no risks associated with urine collection.

#### Risks of mpMRI

Magnetic resonance imaging (MRI) uses a strong magnetic field and radio waves to take pictures of the body. We will obtain pictures of your chest, abdomen and pelvis for this study. The MRI scanner is a metal cylinder surrounded by a strong magnetic field. People are at risk for injury from the MRI magnet if they have some kinds of metal in their body. It may be unsafe for you to

### PATIENT IDENTIFICATION

**Consent to Participate in a Clinical Research Study** 

NIH-2977 (4-17)

File in Section 4: Protocol Consent (1)


have an MRI scan if you have pacemakers or other implanted electrical devices, brain stimulators, some types of dental implants, aneurysm clips (metal clips on the wall of a large artery), metal prostheses (including metal pins and rods, heart valves, and cochlear implants), permanent eyeliner, tattoos, an implanted delivery pump, or shrapnel fragments. Welders and metal workers may have small metal fragments in the eye. You will be screened for these conditions before having any MRI scan. If you have a question about metal in your body, you should inform the staff. You will be asked to complete an MRI screening form before each MRI scan you have.

In addition, all magnetic objects (like watches, coins, jewelry, and credit cards) must be removed before entering the MRI scan room.

People with fear of confined spaces may become anxious during an MRI. Those with back problems may have back pain or discomfort from lying in the scanner. The noise from the scanner is loud enough to damage hearing, especially in people who already have hearing loss. Everyone having a research MRI scan will be fitted with hearing protection. If the hearing protection comes loose during the scan, you should let us know right away.

There are no known long-term risks of MRI scans.

## Risks of gadolinium

During part of the MRI you will receive gadolinium, a contrast agent, through an intravenous (IV) catheter (small tube). It will be done for both research and medical purposes.

The risks of an IV catheter include bleeding, infection, or inflammation of the skin and vein with pain and swelling.

Mild symptoms from gadolinium infusion occur in fewer than 1% of those who receive it and usually go away quickly. Mild symptoms may include coldness in the arm during the injection, a metallic taste, headache, and nausea. In an extremely small number, fewer than one in 300,000 people, more severe symptoms have been reported including shortness of breath, wheezing, hives, and lowering of blood pressure. You should not receive gadolinium if you previously had an allergic reaction to it. You will be asked about such allergic reactions before gadolinium is given.

People with kidney disease are at risk for a serious reaction to gadolinium contrast called "nephrogenic systemic fibrosis (NSF)". This condition always involves the skin and can also involve the muscles, joints, and internal organs. NSF has resulted in a very small number of deaths. A blood test of your kidney function may be done within the month before an MRI scan with gadolinium contrast. You will not receive gadolinium for a research MRI scan if your kidney function is below the safe level.

Most of the gadolinium contrast leaves the body in the urine. However, the FDA has issued a safety alert that indicates small amounts of gadolinium may remain in the body for months to years. The effects of the retained gadolinium are not clear. At this time, retained gadolinium has not been linked to health risks in people whose kidneys work well. Some types of gadolinium contrast drugs are less likely to remain in the body than others. In this study, we will use the gadolinium contrast drugs that are less likely to remain in the body.

Risks of Biopsy

#### PATIENT IDENTIFICATION

Consent to Participate in a Clinical Research Study

NIH-2977 (4-17)

File in Section 4: Protocol Consent (1)


A hollow needle is used to withdraw small cylinders (or cores) of tissue from your tumor using a MRI scan or ultrasound for guidance. The needle is put in 3 to 6 times to get the samples, or cores. This procedure usually causes only brief discomfort at the site from which the biopsy is taken and you will be offered medication to help numb the pain. Biopsy collection may cause bruising and bleeding, but usually does not leave scars. Rarely infection may occur at the needle site.

## Psychological or Social Risks Associated with Loss of Privacy

The following general points are indirectly related to your participation in the research study:

- 1. Unanticipated medical information: During the course of this investigation, it is possible (although not likely) that we will obtain unanticipated information about your health or genetic background.
- 2. Release of genetic information:
- Your privacy is very important to us and we will use many safety measures to protect your privacy. However, in spite of all of the safety measures that we will use, we cannot guarantee that your identity will never become known. Although your genetic information is unique to you, you do share some genetic information with your children, parents, brothers, sisters, and other blood relatives. Consequently, it may be possible that genetic information from them could be used to help identify you. Similarly, it may be possible that genetic information from you could be used to help identify them.
- Patterns of genetic variation also can be used by law enforcement agencies to identify a
  person or his/her blood relatives. Therefore, your genetic information potentially could be
  used in ways that could cause you or your family distress, such as by revealing that you (or
  a blood relative) carry a genetic disease.
- It is possible also that someone could get unauthorized access or break into the system that stores information about you. Every precaution will be taken to minimize this risk.
- There also may be other privacy risks that we have not foreseen.

#### Protections against misuse of genetic information

This study involves genetic testing on samples. Some genetic information can help predict future health problems of you and your family and this information might be of interest to your employers or insurers. The Genetic Information Nondiscrimination Act (GINA) is a federal law that prohibits plans and health insurers from requesting genetic information or using genetic information. It also prohibits employment discrimination based on your health information. However, GINA does not address discrimination by companies that sell life insurance, disability insurance, or long-term care insurance. GINA also does not protect you against discrimination based on an already-diagnosed condition or disease that has a genetic component.

### **Potential Benefits of Participation**

#### Are there benefits to taking part in this study?

The primary aim of this study is to see if mpMRI imaging is a good method to localize and detect prostate cancer. During the study we will also administer 2 drugs in combination. Although these drugs are already approved for treating prostate cancer, less is known about how they work

### PATIENT IDENTIFICATION

### **Consent to Participate in a Clinical Research Study**

NIH-2977 (4-17)

File in Section 4: Protocol Consent (1)


together and what effect they have when given before surgery. It is possible that you will receive some additional personal medical benefit from participating in this trial, but we cannot be certain. These potential benefits could include shrinking of your tumor or lessening of your symptoms, such as pain, that are caused by the cancer. We hope that the knowledge gained from this study may help to detect prostate cancer. We also hope that that you will receive direct benefit to your cancer but because we do not have enough information about how these drugs work together, it is also possible that you may receive no benefit. However, the information gained during this trial may help others with cancer in the future.

## **Alternative Approaches or Treatments**

## What other choices do I have if I do not take part in this study?

Instead of being in this study, you have these options:

- Getting treatment or care for your cancer without being in a study
- Taking part in another study
- Getting comfort care, also called palliative care. This type of care helps reduce pain, tiredness, appetite problems and other problems caused by the cancer. It does not treat the cancer directly. Instead, it tries to improve how you feel. Comfort care tries to keep you as active and comfortable as possible.

Please talk to your doctor about these and other options.

# **Stopping Therapy**

Your doctor may decide to stop your therapy for the following reasons:

- if he/she believes that it is in your best interest
- if you have side effects from the treatment that your doctor thinks are too severe
- if new information shows that another treatment would be better for you

In this case, you will be informed of the reason therapy is being stopped.

You can stop taking part in the study at any time. However, if you decide to stop taking part in the study, we would like you to talk to the study doctor and your regular doctor first.

If you decide at any time to withdraw your consent to participate in the trial, we will not collect any additional medical information about you. However, according to FDA guidelines, information collected on you up to that point may still be provided to Astellas Pharma US Inc or designated representatives. If you withdraw your consent and leave the trial, any samples of yours that have been obtained for the study and stored at the NCI can be destroyed upon request. However, any samples and data generated from the samples that have already been distributed to other researchers or placed in the research databases cannot be recalled and destroyed.

### **Conflict of Interest**

The National Institutes of Health (NIH) reviews NIH staff researchers at least yearly for conflicts of interest. This process is detailed in a Conflict of Interest (COI) Guide. You may ask your research team for a copy of the COI Guide or for more information. Members of the research team

#### PATIENT IDENTIFICATION

Consent to Participate in a Clinical Research Study

NIH-2977 (4-17)

File in Section 4: Protocol Consent (1)


who do not work for NIH are expected to follow these guidelines but they do not need to report their personal finances to the NIH.

No NIH investigator involved in this study receives payments or other benefits from any company whose drug, product or device is being tested.

### Use of Specimens and Data for Future Research

To advance science, it is helpful for researchers to share information they get from studying human samples. They do this by putting it into one or more scientific databases, where it is stored along with information from other studies. A researcher who wants to study the information must apply to the database and be approved. Researchers use specimens and data stored in scientific databases to advance science and learn about health and disease.

We plan to keep some of your specimens and data that we collect and use them for future research and share them with other researchers. We will not contact you to ask about each of these future uses. These specimens and data will be stripped of identifiers such as name, address or account number, so that they may be used for future research on any topic and shared broadly for research purposes. Your specimens and data will be used for research purposes only and will not benefit you. It is also possible that the stored specimens and data may never be used. Results of research done on your specimens and data will not be available to you or your doctor. It might help people who have cancer and other diseases in the future.

If you do not want your stored specimens and data used for future research, please contact us in writing and let us know that you do not want us to use your specimens and/or data. Then any specimens that have not already been used or shared will be destroyed and your data will not be used for future research. However, it may not be possible to withdraw or delete materials or data once they have been shared with other researchers.

### **Genomic Data Sharing**

As part of this research study, we will put your genomic data in a large database for broad sharing with the research community. These databases are commonly called data repositories. The information in this database will include but is not limited to genetic information, race and ethnicity, and sex. If your individual data are placed in one of these repositories, they will be labeled with a code and not with your name or other information that could be used to easily identify you, and only qualified researchers will be able to access them. These researchers must receive prior approval from individuals or committees with authority to determine whether these researchers can access the data.

Summary information about all of the participants included in this study (including you) is being placed in a database and will be available through open access. That means that researchers and non-researchers will be able to access summary information about all the participants included in the study, or summary information combined from multiple studies, without applying for permission. The risk of anyone identifying you with this information is very low.

NIH policies require that genomic data be placed in a repository for sharing. Therefore, we cannot offer you a choice of whether your data will be shared. If you do not wish to have your data placed in a repository, you should not enroll in this study.

#### PATIENT IDENTIFICATION

Consent to Participate in a Clinical Research Study

NIH-2977 (4-17)

File in Section 4: Protocol Consent (1)


#### **PAYMENT**

## Will you receive any type of payment for taking part in this study?

You will not receive any payment for taking part in this study.

#### REIMBURSEMENT

# Will you receive reimbursement or direct payment by NIH as part of your participation?

On this study, the NCI will reimburse the cost for some of your expenses such as those for hotel, travel, meals. Some of these costs may be paid directly by the NIH and some may be reimbursed after you have paid. The amount and form of these payments are determined by the NCI Travel and Lodging Reimbursement Policy. You will be given a summary of the policy which provides more information.

If your travel to the NIH Clinical Center (e.g. flight, hotel) is arranged and paid for by the NIH, the agency making the reservations and their representatives will have access to your identifiable information.

#### COSTS

## Will taking part in this research study cost you anything?

NIH does not bill health insurance companies or participants for any research or related clinical care that you receive at the NIH Clinical Center.

- You will receive study treatment at no charge to you. This may include surgery, medicines, laboratory testing, or scans done at the Clinical Center, National Institutes of Health (NIH), or arranged for you by the research team to be done outside the Clinical Center, NIH if the study related treatment is not available at the NIH.
- There are limited funds available to cover the cost of some tests and procedures performed outside the Clinical Center, NIH. You may have to pay for these costs if they are not covered by your insurance company.
- Medicines that are not part of the study treatment will not be provided or paid for by the Clinical Center. NIH.
- Once you have completed taking part in the study, medical care will no longer be provided by the Clinical Center, NIH.

### CLINICAL TRIAL REGISTRATION AND RESULTS REPORTING

A description of this clinical trial will be available on <a href="http://www.ClinicalTrials.gov">http://www.ClinicalTrials.gov</a>, as required by U.S. Law. This Web site will not include information that can identify you. At most, the Web site will include a summary of the results. You can search this Web site at any time.

### CONFIDENTIALITY PROTECTIONS PROVIDED IN THIS STUDY

### Will your medical information be kept private?

We will do our best to make sure that the personal information in your medical record will be kept private. However, we cannot guarantee total privacy. Organizations that may look at and/or copy your medical records for research, quality assurance, and data analysis include:

#### PATIENT IDENTIFICATION

### **Consent to Participate in a Clinical Research Study**

NIH-2977 (4-17)

File in Section 4: Protocol Consent (1)


- The NIH and other government agencies, like the Food and Drug Administration (FDA), which are involved in keeping research safe for people.
- National Institutes of Health Intramural Institutional Review Board

The researchers conducting this study and the NIH follow applicable laws and policies to keep your identifying information private to the extent possible. However, there is always a chance that, despite our best efforts, your identity and/or information about your participation in this research may be inadvertently released or improperly accessed by unauthorized persons.

In most cases, the NIH will not release any identifiable information collected about you without your written permission. However, your information may be shared as described in the section of this document on sharing of specimens and data, and as further outlined in the following sections.

Further, the information collected for this study is protected by NIH under a Certificate of Confidentiality and the Privacy Act.

# **Certificate of Confidentiality**

To help us protect your privacy, the NIH Intramural Program has received a Certificate of Confidentiality (Certificate). With this certificate, researchers may not release or use data or information about you except in certain circumstances.

NIH researchers must not share information that may identify you in any federal, state, or local civil, criminal, administrative, legislative, or other proceedings, for example, if requested by a court.

The Certificate does not protect your information when it:

- 1. is disclosed to people connected with the research, for example, information may be used for auditing or program evaluation internally by the NIH; or
- 2. is required to be disclosed by Federal, State, or local laws, for example, when information must be disclosed to meet the legal requirements of the federal Food and Drug Administration (FDA);
- 3. is for other research;
- 4. is disclosed with your consent.

The Certificate does not prevent you from voluntarily releasing information about yourself or your involvement in this research.

The Certificate will not be used to prevent disclosure to state or local authorities of harm to self or others including, for example, child abuse and neglect, and by signing below you consent to those disclosures. Other permissions for release may be made by signing NIH forms, such as the Notice and Acknowledgement of Information Practices consent.

### **Privacy Act**

The Federal Privacy Act generally protects the confidentiality of your NIH medical records we collect under the authority of the Public Health Service Act. In some cases, the Privacy Act protections differ from the Certificate of Confidentiality. For example, sometimes the Privacy Act allows release of information from your medical record without your permission, for example, if it is requested by Congress. Information may also be released for certain research purposes with due consideration and protection, to those engaged by the agency for research purposes, to certain

### PATIENT IDENTIFICATION

Consent to Participate in a Clinical Research Study

NIH-2977 (4-17)

File in Section 4: Protocol Consent (1)


federal and state agencies, for HIV partner notification, for infectious disease or abuse or neglect reporting, to tumor registries, for quality assessment and medical audits, or when the NIH is involved in a lawsuit. However, NIH will only release information from your medical record if it is permitted by both the Certificate of Confidentiality and the Privacy Act.

#### POLICY REGARDING RESEARCH-RELATED INJURIES

The NIH Clinical Center will provide short-term medical care for any injury resulting from your participation in research here. In general, no long-term medical care or financial compensation for research-related injuries will be provided by the NIH, the NIH Clinical Center, or the Federal Government. However, you have the right to pursue legal remedy if you believe that your injury justifies such action.

### PROBLEMS OR QUESTIONS

If you have any problems or questions about this study, or about your rights as a research participant, or about any research-related injury, contact the Principal Investigator, Fatima Karzai, <a href="mailto:fatima.karzai@nih.gov">fatima.karzai@nih.gov</a>, at 301-480-7174. You may also call the NIH Clinical Center Patient Representative at 301-496-2626, or the NIH Office of IRB Operations at 301-402-3713, if you have a research-related complaint or concern.

### CONSENT DOCUMENT

Please keep a copy of this document in case you want to read it again.

NIH-2977 (4-17)

File in Section 4: Protocol Consent (1)


| to discuss it and to ask question | ns. I consent to participate in this study. | d have been given the opportun |
|---|---|---|
| Signature of Research Participa | ant Print Name of Research Pa | nrticipant Date |
| about this study and have been to make research decisions on b | ntative (LAR) for an Adult Unable to Consequence of given the opportunity to discuss it and to ask obehalf of the adult participant unable to consent cable, the information in the above consent was to participate in the study. | questions. I am legally authoriz<br>t and have the authority to provi |
| Signature of LAR | Print Name of LAR | Date |
| Investigator: | | |
| Signature of Investigator | Print Name of Investigator | Date |
| Signature of Witness* | Print Name of Witness | |
| orginature or withess | Time Ivalie of Witness | Date |
| *NIH ADMINISTRATIVE | SECTION TO BE COMPLETED REG | |
| INTERPRETER: | | |
| INTERPRETER: An interpreter, or other inc | dividual, who speaks English and the participand consent and served as a witness. The investi | nt's preferred language facilita |
| An interpreter, or other income also serve as the witness. An interpreter, or other income also serve as the witness. | dividual, who speaks English and the participal consent and served as a witness. The investigation of the dividual, who speaks English and the participal consent but did not serve as a witness. The na | nt's preferred language facilitating consent may not be supported to the person of the person |
| INTERPRETER: An interpreter, or other income also serve as the witness. An interpreter, or other income also serve as the witness. | dividual, who speaks English and the participand consent and served as a witness. The investigation of the participand consent but did not serve as a witness. The national consent but did not serve as a witness. | nt's preferred language facilita<br>igator obtaining consent may<br>nt's preferred language facilita<br>ame or ID code of the person |


IRB APPROVAL DATE: 05/18/2022